CLINICAL TRIAL: NCT03220334
Title: Healing Effects of Autologous Platelet Rich Plasma on Gastric Ulcer Caused by Endoscopic Submucosal Dissection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, YooJin Lee, Assistant professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12-181
Record Dates: First submitted 2017-07-09; First posted 2017-07-18 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Platelet-rich Plasma; Endoscopic Submucosal Dissection
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apply platelet rich plasma to the artificial gastric ulcer (Experimental)
  Interventions: Drug: Platelet rich plasma
- Apply normal saline to the artificial gastric ulcer (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Platelet rich plasma — The experimental group was treated with PRP for artificial gastric ulcer after ESD.
  Other Names: PRP
  Arms: Apply platelet rich plasma to the artificial gastric ulcer
Drug: Normal saline — The control group was treated with normal saline for artificial gastric ulcer after ESD.
  Arms: Apply normal saline to the artificial gastric ulcer

SUMMARY:
In Korea, where the prevalence of gastric tumors is high, the use of ESD as a treatment for gastric cancer will continue to increase. Considering that there are no special measures to prevent side effects (bleeding, perforation, etc.) of this procedure, it is possible to reduce the large medical costs through the discovery of substances that can promote gastric mucosal healing. Mechanism of PRP-based materials in the regeneration of gastric mucosal damage can be used to understand the pathophysiology of ulcers. In the future, it can be suggested as a new treatment for gastrointestinal tract damage such as intractable ulcer, perforation, mucosal fistula, gastrointestinal bleeding caused by esophagus, small intestine and large intestine as well as ulcer treatment by endoscopic procedure.

DETAILED DESCRIPTION:
Background:In Korea, where the prevalence of gastric tumors is high, the use of ESD as a treatment for gastric cancer will continue to increase. Considering that there are no special measures to prevent side effects (bleeding, perforation, etc.) of this procedure, it is possible to reduce the large medical costs through the discovery of substances that can promote gastric mucosal healing. Platelet-rich plasma (PRP) has demonstrated efficacy in preclinical endoscopic resection models.

Aim: Evaluate the efficacy of PRP on participants submitted to ESD.

Material and Methods: The investigators have evaluated a prospective clinical study. The investigators have included 10 participants submitted to ESD. Patients were informed and accepted to participate with a written consent. Prior to endoscopy PRP was obtained from autologous blood with a commercial kit. Resection was performed with standard technique. Immediately after the procedure, autologous PRP is applied to the artificial gastric ulcer using endoscopic spray. Participants were followed-up after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopic lesion submitted to endoscopic resection (ESD)

Exclusion Criteria:

* Ineligibility to endoscopic resection
* Patients who declined to participate in this study
* Patients who had hematologic diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Recovery of artificial gastric ulcer | 2 weeks
  Measure the ulcer size with an endoscopy.

SECONDARY OUTCOMES:
Recovery of artificial gastric ulcer | 4 weeks
  Measure the ulcer size with an endoscopy.
Occurrence of postprocedure complication | 2 weeks
  Postprocedure complications were investigated by patient examination and endoscopy.
Occurrence of postprocedure complication | 4 weeks
  Postprocedure complications were investigated by patient examination and endoscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- KeimyungUniversity, Daegu, Jung-gu, South Korea